CLINICAL TRIAL: NCT07049094
Title: A Multicenter, Single-blind, Randomized Controlled Study on the Analgesic Effect of Scalp Nerve Block Using Bupivacaine Liposomes for Postoperative Pain Relief After Craniotomy
Brief Title: The Analgesic Effect of Scalp Nerve Block Using Bupivacaine Liposomes for Postoperative Pain Relief After Craniotomy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Diansan Su, Chair of the Department of Anesthesiology, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZJU2025B0536
Record Dates: First submitted 2025-06-08; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Brain Tumor Adult; Cerebrovascular Disease
Keywords: supratentorial craniotomy; postoperative analgesia
MeSH Terms: conditions — Cerebrovascular Disorders | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- scalp nerve block with 0.25% hydrochloride bupivacaine and 0.67% bupivacaine liposome solution (Experimental): In this group, patients use 0.25% hydrochloride bupivacaine and 0.67% bupivacaine liposome solution for scalp nerve block
  Interventions: Drug: scalp nerve block with 0.25% hydrochloride bupivacaine and 0.67% bupivacaine liposome solution
- scalp nerve block with 0.50% hydrochloride bupivacaine (Active Comparator): In this group, patients use 0.50% hydrochloride bupivacaine for scalp nerve block
  Interventions: Drug: scalp nerve block with 0.50% hydrochloride bupivacaine

INTERVENTIONS:
Drug: scalp nerve block with 0.25% hydrochloride bupivacaine and 0.67% bupivacaine liposome solution — Using 0.25% hydrochloride bupivacaine and 0.67% bupivacaine liposome solution for scalp nerve block
  Arms: scalp nerve block with 0.25% hydrochloride bupivacaine and 0.67% bupivacaine liposome solution
Drug: scalp nerve block with 0.50% hydrochloride bupivacaine — Using 0.50% hydrochloride bupivacaine for scalp nerve block
  Arms: scalp nerve block with 0.50% hydrochloride bupivacaine

SUMMARY:
After undergoing craniotomy, 60% to 84% of neurosurgery patients experience moderate to severe acute pain, primarily in the first 48 hours. This pain is mostly superficial, affecting the muscles and soft tissues around the skull. Poor pain management can lead to complications such as restlessness, nausea, hypertension, increased intracranial pressure, and prolonged recovery, potentially resulting in chronic headaches.

Opioids are commonly used to manage this pain but can cause significant side effects like sedation, nausea, and increased intracranial pressure, which can mask serious conditions. Non-opioid medications and scalp infiltration techniques can help but may not provide sufficient pain relief for the duration needed.

Currently, multimodal analgesia, particularly scalp nerve blocks, is advocated in neurosurgical recovery practices. These blocks are effective and simpler to perform, but the effects of long-acting local anesthetics, like bupivacaine, typically last only 24 hours. Since pain often persists longer than that, there is a need for better pain management strategies.

Liposome bupivacaine is a new long-acting local anesthetic approved by the FDA, offering pain relief for up to 72 hours compared to regular bupivacaine's 8-hour duration. Its effectiveness has been confirmed in various nerve block procedures, but it has not been reported for scalp nerve blocks. This study aims to investigate whether liposome bupivacaine scalp nerve blocks can provide long-lasting postoperative pain relief, promote quicker recovery, and reduce complications in neurosurgery patients.

DETAILED DESCRIPTION:
This study aims to compare the analgesic efficacy and safety of hydrochloride bupivacaine versus liposomal bupivacaine in patients undergoing elective cranial surgery. The protocol is designed to rigorously assess pain management outcomes, recovery quality, and potential complications through a randomized, single-blind, controlled trial.

Study Design and Methodology After a comprehensive screening process, eligible patients are randomized into two groups: the control group receiving hydrochloride bupivacaine and the experimental group receiving a combination of hydrochloride bupivacaine and liposomal bupivacaine. Randomization was implemented using a pre-generated data list to ensure allocation concealment and minimize selection bias. The single-blind design ensures that patients are unaware of their group assignment, while clinicians administering the drugs are informed to ensure proper preparation and delivery.

Preoperative Assessment

Prior to surgery, all subjects undergo a thorough evaluation, including:

1. Neurological Assessment: Consciousness levels are assessed using the Glasgow Coma Scale (GCS).
2. Laboratory Testing: Electrocardiograms, routine blood tests (e.g., RBC, WBC, hemoglobin, platelet count), and liver/kidney function tests (e.g., ALT, AST, serum creatinine, BUN) are performed to confirm eligibility and detect any underlying conditions.
3. Pain and Recovery Familiarization： Patients are introduced to the Numeric Rating Scale (NRS) for pain, the Objective Pain Assessment Scale (OBAS), and the Quality of Recovery-15 (QoR15) scale to standardize postoperative data collection.

Anesthesia and Intraoperative Protocol Upon admission to the operating room, inclusion/exclusion criteria are re-evaluated, and baseline vitals (SPO2, BP, ECG) are monitored. Peripheral intravenous and arterial lines are established for drug administration and invasive blood pressure monitoring.

1. General Anesthesia Induction:

   Induction agents include midazolam/remimazolam, propofol, sufentanil, and rocuronium/cisatracurium.

   Endotracheal intubation is performed after 3 minutes of induction, followed by mechanical ventilation with a tidal volume of 6-8 ml/kg and a respiratory rate of 10-12 breaths/min to maintain end-tidal CO2 at 30-40 mmHg.
2. Maintenance of Anesthesia:

   Anesthesia is maintained with sevoflurane, propofol, remifentanil, and either cisatracurium or rocuronium.

   Dexamethasone (5 mg) and betamethasone (4 mg) are routinely administered during induction to reduce inflammation and nausea.

   To avoid confounding variables, non-steroidal anti-inflammatory drugs, additional opioids (e.g., dezocine, norfentanyl), and dexmedetomidine are excluded.
3. Scalp Nerve Blocks： Scalp nerve blocks are performed bilaterally before the surgical incision to enhance analgesia. The blocks target six major nerve groups (e.g., superior orbital, supraorbital, zygomatic-temporal, auriculotemporal, greater occipital, and lesser occipital nerves) using precise anatomical landmarks and standardized volumes of local anesthetic.

Drug Preparation and Administration Control Group: 20 ml of 0.75% hydrochloride bupivacaine is diluted with 10 ml saline and divided into three 10 ml doses.

Experimental Group: 10 ml of 0.75% hydrochloride bupivacaine is mixed with 15 ml of 1.33% liposomal bupivacaine and 5 ml saline, also divided into three 10 ml doses.

The prepared solutions are administered during nerve blocks under aseptic conditions.

Recovery and Extubation Postoperatively, sedatives are discontinued, and muscle relaxation is reversed with either neostigmine (1-2 mg) and atropine (0.5-1 mg) or sugammadex (2 mg/kg). Extubation is performed when patients achieve a score of >9 on Godet et al.'s scoring criteria. Patients are monitored in the Post-Anesthesia Care Unit (PACU) for 1 hour.

Postoperative Rescue Analgesia Rescue analgesia is provided if NRS scores are ≥4, with intravenous non-steroidal anti-inflammatory drugs or other clinically appropriate interventions. All rescue analgesia events are documented.

Measures to Minimize Bias Randomization: Ensures equal distribution of confounding factors between groups.

Blinding: Subjects are blinded to their group assignment to reduce placebo effects.

Standardized Assessment Tools: NRS, OBAS, and QoR15 scales are used to objectively evaluate pain and recovery outcomes.

Clinical Indicator Assessment

Primary and secondary outcomes are measured at predefined postoperative time points:

Primary Endpoint: Resting AUC-NRS scores within 48 hours postoperatively (PACU discharge, 4 hours post-op, 8 hours post-op, and on POD1 at 8:30, 12:00, and 16:00).

Secondary Endpoints:

Coughing AUC-NRS scores within 48 hours postoperatively. Resting NRS scores at PACU discharge and on POD1-3. OBAS scores, QoR15 scores, and incidence of postoperative complications (e.g., nausea, vomiting, nerve block-related issues).

Subject Selection and Withdrawal Detailed inclusion and exclusion criteria ensure the recruitment of a homogenous study population. Subjects may withdraw at any time, and procedures are in place to document and address missed visits and loss to follow-up.

Sample Size and Statistical Power A total of 218 subjects are required to achieve adequate statistical power, accounting for potential dropouts. This sample size is calculated based on the primary endpoint to detect clinically significant differences between groups.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* ASA I-III
* Scheduled for elective cranial surgery
* Informed consent from the patient or legal representative

Exclusion Criteria:

* Preoperative Glasgow score < 15
* Preoperative headache with NRS ≥ 4
* Anticipated postoperative sedation or extubation difficulties requiring mechanical ventilation
* Inability to understand the numerical rating scale (NRS)
* Allergies or contraindications to amide local anesthetics, opioids, or NSAIDs
* Long-term opioid or corticosteroid treatment (> 2 weeks)
* History of drug abuse in the past 2 years
* Daily alcohol consumption exceeding 3 standard doses
* Mental or cognitive disorders affecting perioperative assessment
* Contraindications for nerve blocks, including infection or tumors at the puncture site, diagnosed diabetic peripheral neuropathy, or inability to cooperate
* Severe liver dysfunction (Child-Pugh class C), severe renal dysfunction (requiring dialysis preoperatively), or severe heart failure (METS < 4)
* Pregnant or breastfeeding women
* History of craniotomy or pre-existing pathological pain conditions (e.g., migraines, trigeminal neuralgia)
* Incisions for craniotomy extending beyond the area covered by the scalp nerve blocks
* Participation in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2025-06-25 (Estimated); Primary Completion 2027-06-25 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Resting Area Under the Curve - Numerical Rating Scale score within 48 hours after surgery | 2 hours post-operation, 4 hours post-operation, 8 hours post-operation, postoperative day 1 8:30, postoperative day 12:00, postoperative day 1 16:00
  The Numerical Rating Scale (NRS) is a widely used tool for assessing the intensity of pain. It is a self-reported scale where patients are asked to rate their pain on a numerical scale ranging from 0 to 10.
  Minimum Value (0): Indicates "No Pain" or the complete absence of pain. This is the best possible outcome for the patient.
  Maximum Value (10): Indicates "Worst Pain Imaginable" or the most severe pain the patient can conceive. This is the worst possible outcome for the patient.

SECONDARY OUTCOMES:
Area Under the Curve - Numerical Rating Scale score during coughing within 48 hours after surgery | within 48 hours after surgery
  The Numerical Rating Scale (NRS) is a widely used tool for assessing the intensity of pain. It is a self-reported scale where patients are asked to rate their pain on a numerical scale ranging from 0 to 10.
  Minimum Value (0): Indicates "No Pain" or the complete absence of pain. This is the best possible outcome for the patient.
  Maximum Value (10): Indicates "Worst Pain Imaginable" or the most severe pain the patient can conceive. This is the worst possible outcome for the patient.
Numerical Rating Scale score at rest after discharge from Post-Anesthesia Care Unit on Postoperative Day 1 to Day 3 | Postoperative Day 1 to Day 3
  The Numerical Rating Scale (NRS) is a widely used tool for assessing the intensity of pain. It is a self-reported scale where patients are asked to rate their pain on a numerical scale ranging from 0 to 10.
  Minimum Value (0): Indicates "No Pain" or the complete absence of pain. This is the best possible outcome for the patient.
  Maximum Value (10): Indicates "Worst Pain Imaginable" or the most severe pain the patient can conceive. This is the worst possible outcome for the patient.
Numerical Rating Scale score during coughing after discharge from Post-Anesthesia Care Unit on Postoperative Day 1 to Postoperative Day 3 | Postoperative Day 1 to Day 3
  The Numerical Rating Scale (NRS) is a widely used tool for assessing the intensity of pain. It is a self-reported scale where patients are asked to rate their pain on a numerical scale ranging from 0 to 10.
  Minimum Value (0): Indicates "No Pain" or the complete absence of pain. This is the best possible outcome for the patient.
  Maximum Value (10): Indicates "Worst Pain Imaginable" or the most severe pain the patient can conceive. This is the worst possible outcome for the patient.
Analgesic use within 48 hours after surgery | within 48 hours after surgery
Overall Benefit Assessment Score for Analgesia within 48 Hours after Surgery | within 48 Hours after Surgery
  The Numerical Rating Scale (NRS) is a widely used tool for assessing the intensity of pain. It is a self-reported scale where patients are asked to rate their pain on a numerical scale ranging from 0 to 10.
  Minimum Value (0): Indicates "No Pain" or the complete absence of pain. This is the best possible outcome for the patient.
  Maximum Value (10): Indicates "Worst Pain Imaginable" or the most severe pain the patient can conceive. This is the worst possible outcome for the patient.
Postoperative Day 5 Quality of Recovery (Quality of Recovery 15) | Postoperative Day 5
  The QoR-15 consists of 15 items across five dimensions: physical comfort, emotional state, physical independence, psychological support, and pain. Patients are asked to score each item on a numeric scale (e.g., 0-10), where higher scores reflect better recovery. This self-reported questionnaire provides a comprehensive measure of the patient's postoperative recovery experience by addressing both subjective and objective aspects of well-being.
  In summary:
  Goal: To assess the quality of recovery on the fifth postoperative day. Measurement Tool: QoR-15 questionnaire. Domains Assessed: Physical comfort, emotional state, physical independence, support from others, and pain management.
Nausea and Vomiting within 48 Hours after Surgery | within 48 Hours after Surgery
  Number of Participants Experiencing Nausea and Vomiting within 48 Hours after Surgery

OTHER OUTCOMES:
Monitoring postoperative adverse events according to the Common Terminology Criteria for Adverse Events version 5.0 | postoperative day 1 to day 5
Infection and bleeding at the puncture site | postoperative day1 to day5
complications of scalp nerve block (ptosis, shallow nasolabial fold, facial asymmetry, speech with air leakage, salivation) | postoperative day1 to day5

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided